CLINICAL TRIAL: NCT05430425
Title: Comparison of the Efficiency of Classical and I-GEL LMAs Selected by Different Methods in Providing a Safe Airway
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Yunus Emre (Other)
Responsible Party: Sponsor-Investigator, Yunus Emre, SPECIALIST DOCTOR, Ankara Training and Research Hospital
Organization: Ankara Training and Research Hospital (Other)
Other Study IDs: ytuncdemir-lma
Record Dates: First submitted 2022-06-13; First posted 2022-06-24 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Airway Complication of Anesthesia
Keywords: anesthesia; laryngeal mask; safe respiratory tract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- body weight: (grup VA; igel=n:40 clasic lma n=40),
  Interventions: Other: respiratory safety
- thyromental distance: grup T; igel=n:40 clasic lma n=40)
  Interventions: Other: respiratory safety
- resize with 3 fingers: grup p; igel=n:40 clasic lma n=40
  Interventions: Other: respiratory safety

INTERVENTIONS:
Other: respiratory safety — Which of the 3 lma selection methods is effective in ensuring respiratory safety?

SUMMARY:
In recent years, the use of laryngeal masks has been increasing in operating room and non-operating room anesthesia applications. Patients with inappropriate LMA may develop high leakages, gastric distension and inadequate ventilation during ventilation. If the laryngeal masks used to provide a safe airway in the patient are not selected in the appropriate size, adequate ventilation may not be provided, which may lead to various complications such as increased morbidity and mortality. In order to prevent and predict the bad results that may occur, we foresee which method can be chosen more appropriately for the patients and will guide the clinicians.

DETAILED DESCRIPTION:
The laryngeal mask (LMA) is a subragglottic airway device commonly used to provide lung ventilation during general anesthesia. In this study, we aimed to compare the efficacy of classical and I-GEL LMA selected with different techniques.

Successful placement of the Laryngeal Mask Airway (LMA) largely depends on the correct size selection.

The size of the laryngeal mask airway is usually determined by the weight of the patient. However, in some cases an alternative method can be used. The weight of the patient is sometimes unknown (eg, obese, malnourished, sedentary or unconscious patients) and can be unpredictable, especially in children. Therefore, it will be useful to have alternative ways (according to 1. body weight, 2. thyromental distance, 3. dimensioning with three fingers) in determining the appropriate size of the laryngeal mask size. These different methods should be simple to perform and easy to remember.

LMA is increasingly used in elective surgery, resuscitation, difficult airway and emergency situations. Successful use of the LMA largely depends on the correct size selection, method of insertion, and cuff sealing. Placing an improperly sized LMA can result in incorrect positioning and incorrect ventilation

ELIGIBILITY:
Inclusion Criteria:

* Elective cases between the ages of 18-65,
* ASA I-II,
* who will be fitted with an LMA by the anesthesia clinic,
* and whose consent has been obtained

Exclusion Criteria:

->65 years old,

* excessive cachectic or body mass index (BMI) >30 kg/m2,
* those with high risk of regurgitation or aspiration (large hiatal hernia, Zenker's diverticulum, scleroderma, pregnancy, history of gastroesophageal reflux disease, uncontrolled diabetes mellitus and obesity),
* potentially difficult airway (history of airway difficulty, mouth opening <2 cm,
* Mallampati class 4,
* limited neck extension or cervical spine pathology),
* airway pathology,
* decreased presence of pulmonary or chest wall compliance,
* preoperative sore throat,
* planned operation Patients with a duration of >2 hours and who need a prone position during surgery will not be included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases aged between 18-65 years, whose elective consents have been obtained, and who will be placed under ASA I-II and LMA under general anesthesia will be included.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-06-22 (Estimated); Primary Completion 2022-08-07 (Estimated); Study Completion 2022-10-22 (Estimated)

PRIMARY OUTCOMES:
Selection of the appropriate supraglottic airway device for the patient | three month
  selecting the most appropriate laryngeal mask to ensure a safe airway. laryngeal mask; It can be selected according to body weight, thyromental distance and three finger size of the hand.Among these mask selection methods, the mask with the best effectiveness and the least complication will be selected

IPD SHARING:
Plan to Share IPD: Undecided